CLINICAL TRIAL: NCT06744413
Title: Prehabilitation to Improve Heart Rate Variability In Surgical Cancer Patients: a randoMized controllEd Trial
Brief Title: Prehabilitation to Improve Heart Rate Variability (PRIME)
Acronym: PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Dott. Fabio Guarracino (Unknown); Prof. Gilda Cinnella (Unknown); Dott. Filippo Sanfilippo (Unknown)
Responsible Party: Principal Investigator, Giovanni Landoni, Full professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PNRR-MCNT2-2023-12377934
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cancer Surgery
Keywords: Cancer surgery; Prehabilitation; Multimodal prehabilitation program; Standard care treatment; Hospital stay; Functional walking; Nutrition; Diet; Exercise; Relaxation; Functional recovery; Anesthesiology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Prehabilitation arm groups will receive preoperative intervention which includes exercise training, nutritional therapy and anxiety reducing techniques, aimed at preventing or attenuating surgery-driven functional decline.
  Interventions: Behavioral: Multimodal prehabilitation program
- Control group (No Intervention): Standard care treatment: application of ERAS pathways (Enhanced Recovery After Surgery)

INTERVENTIONS:
Behavioral: Multimodal prehabilitation program — A tailored intervention will be prescribed if specific physical, nutritional or psychological impairments will be identified during the assessment phase. Based on the data obtained during the multimodal assessment, different domains and levels of care will be prescribed, focusing on exercise training, and/or nutrition optimization, and/or distress-coping techniques. Different combinations of these three domains will be utilized to maximize their synergistic anabolic effect.
  The duration of the program will be set at 4 weeks.
  Arms: Prehabilitation

SUMMARY:
Cancer patients require chronic management and care. For those individuals living with cancer, a comprehensive approach that acknowledges the interdisciplinary nature of their condition can help guide appropriate care strategies and support their overall well-being. Approximately 45% of patients diagnosed with cancer undergo surgery to remove their tumor. Despite the advancements in surgical techniques, anesthesia, and perioperative care, major cancer surgeries still pose a significant challenge leading to a considerable decline in physiological and functional capacity. Traditionally, efforts focused on postoperative rehabilitation to enhance recovery. Recently, prehabilitation, a form of rehabilitation which aims to improve functional capacity before surgery, has gained attention for its potential benefits in improving surgical outcomes. However, prehabilitation lacks objective assessment measures to evaluate its effectiveness. Developing validated outcome measures is essential to enhance the impact of prehabilitation on surgical outcomes and long-term care for cancer patients. Heart rate variability (HRV) is a physiological parameter that measures the variation in time intervals between consecutive heartbeats, reflecting the autonomic nervous system activity which might serve as a valuable solution for objective outcome measures in evaluating the effectiveness of prehabilitation for cancer patients, providing an objective tool to assess and monitor physiological response to stress, recovery capacity, and autonomic nervous system activity. A multicenter randomized controlled trial will be conducted to assess the impact of a multimodal prehabilitation program on HRV. Patients aged 18 or older, scheduled for elective major cancer surgery will be randomized to receive either prehabilitation or standard care. The prehabilitation arm will receive a program involving home-based physical, nutritional, and psychological interventions for at least four weeks. Participants allocated to the control group will receive usual care. Patients will be followed throughout the study using an innovative mobile application, allowing for real-time monitoring and data collection during the prehabilitation program. The study has two primary outcomes: A) to assess the impact of prehabilitation on increasing preoperative HRV in chronic cancer patients undergoing surgery; B) to assess the effect of prehabilitation on length of hospital stay.

DETAILED DESCRIPTION:
Cancer patients require long-term management and ongoing care due to the chronic nature of their condition. Major cancer surgeries pose significant challenges, resulting in a decline in physiological and functional capacity. Traditionally, postoperative rehabilitation has been the most suitable intervention to improve functional recovery. Prehabilitation, which aims to enhance patients' functional capacity before surgery and to improve patients' ability to cope with physiological stress, is considered the best form of rehabilitation. Through multimodal strategies like exercise, nutrition and psychological support, prehabilitation can improve surgical outcomes for cancer patients. However, prehabilitation lacks objective assessment measures. Heart rate variability (HRV), a physiological parameter measuring variation in heartbeats, reflects autonomic nervous system activity and an increase in HRV is associated with fitness and recovery capacity in sports medicine. Psychological factors, nutritional status and physical exercise influence HRV. Hence, HRV could be used to objectively assess prehabilitation interventions. In addition, HRV is widely used in risk assessment in cardiology, and a reduction in HRV is recognized to be associated with complications and mortality. Despite its evident potential in risk assessment, HRV has never been utilized in preoperative assessments.

This is an international, multicenter, parallel-group, randomized study in chronic cancer patients undergoing surgery. Adult men and women patients who are eligible according to the inclusion/exclusion criteria will be randomized to study the effect of prehabilitation versus standard care on heart rate variability (HRV).

A total of 600 patients will be recruited by systematic screening of patients scheduled for elective surgical procedures. All patients undergoing major cancer surgery will be screened for eligibility and those who meet the inclusion/exclusion criteria will be approached for consent. Research personnel will use a web-based randomization system to assign patients (1:1 ratio) to either the prehabilitation or control arm. Study personnel will also collect data on recruitment rates, with reasons for non-enrollment.

Eligible patients will be randomly assigned to one of two treatments:

1. Multimodal prehabilitation program for four weeks starting as soon as possible before surgery;
2. Standard care.

The multimodal prehabilitation program will be individualized by carefully integrating and adapting various components to meet individual needs. The program will last four weeks (plus maintenance in case of delayed surgery), and will incorporate exercise training, nutritional therapy, and anxiety reduction techniques. After enrollment, patients will receive initial contact from trained personnel through telemedicine. To ensure personalized care, a comprehensive assessment will be conducted to identify specific physical, nutritional, or psychological challenges. Based on this assessment, a customized intervention plan will be prescribed to achieve tailored exercise training, optimized nutrition, and effective distress-coping strategies. Patients will be requested to download a dedicated smartphone application, which will comprehensively monitor and track their progress towards achieving their prehabilitation goals. After completing the four-week program, patients will continue a maintenance program until surgery.

The first HRV measurement will be performed for 5 minutes in an isolated room, after signing the written consent and before randomization, on the day of screening which occurs several weeks before surgery. The second HRV measurement will be performed the day before surgery. Both HRV time-domain measurements and HRV frequency-domain measurements will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo elective major abdominal or thoracic cancer surgery;
2. Scheduled to undergo surgery at least three weeks after enrollment;
3. Age ≥ 18 years;
4. Provide written informed consent;
5. Willing and able to use smartphone application.

Exclusion Criteria:

1. Presenting with very poor functional capacity;
2. American Society of Anesthesiologists (ASA) physical status classes 5-6;
3. Disabling orthopedic, neuromuscular, and psychiatric diseases or other conditions that preclude participation in a prehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Assess the impact of prehabilitation on heart rate variability | Preoperative
  This primary outcome measure will be the change in the standard deviation of normal-to-normal intervals (SDNN) from baseline to the day before surgery.
Days at home within first 30 days after surgery | 30-days after surgery
  The mean number of days at home in the first 30 days after surgery will be compared between groups

SECONDARY OUTCOMES:
Quality of life at 30 days | 30-days after surgery
  Assess quality of life in the first 30 days at home after surgery using the EuroQol-5 Dimension (EQ-5D-5L) questionnaire, a validated tool for evaluating health-related quality of life. The outcome will be reported as the mean EQ-5D-5L index score and the mean EQ-VAS score measured at 30 days postoperatively.
30-days postoperative complication | 30-days after surgery
  Assess the occurrence of postoperative complications in the first 30 days after surgery
Correlation between preoperative standard deviation of all normal to normal R-R intervals (SDNN) and quality of life at 30 days postoperatively | 30-days after surgery
  Investigate the association between preoperative heart rate variability (HRV) and life at 30 days postoperatively
Correlation between preoperative SDNN and DAH-30 | 30-days after surgery
  Investigate the association between preoperative heart rate variability (HRV) and the days alive and at home within 30 days after surgery (DAH-30)
Correlation between preoperative SDNN and postoperative complication | 30-days after surgery
  Investigate the association between preoperative heart rate variability (HRV) and postoperative complication

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Guarracino, Doctor, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (4):
- Italy (4):
  - Azienda Ospedaliero Universitaria Policlinico San Marco di Catania, Catania
  - Università di Foggia, Foggia
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The Atherosclerosis Risk in Communities (ARIC) Study: design and objectives. The ARIC investigators. Am J Epidemiol. 1989 Apr;129(4):687-702. PMID 2646917
- [Background] Zhou X, Ma Z, Zhang L, Zhou S, Wang J, Wang B, Fu W. Heart rate variability in the prediction of survival in patients with cancer: A systematic review and meta-analysis. J Psychosom Res. 2016 Oct;89:20-5. doi: 10.1016/j.jpsychores.2016.08.004. Epub 2016 Aug 8. PMID 27663106
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Scheede-Bergdahl C, Minnella EM, Carli F. Multi-modal prehabilitation: addressing the why, when, what, how, who and where next? Anaesthesia. 2019 Jan;74 Suppl 1:20-26. doi: 10.1111/anae.14505. PMID 30604416
- [Background] Orange ST, Northgraves MJ, Marshall P, Madden LA, Vince RV. Exercise prehabilitation in elective intra-cavity surgery: A role within the ERAS pathway? A narrative review. Int J Surg. 2018 Aug;56:328-333. doi: 10.1016/j.ijsu.2018.04.054. Epub 2018 May 3. PMID 29730070
- [Background] Nolan J, Batin PD, Andrews R, Lindsay SJ, Brooksby P, Mullen M, Baig W, Flapan AD, Cowley A, Prescott RJ, Neilson JM, Fox KA. Prospective study of heart rate variability and mortality in chronic heart failure: results of the United Kingdom heart failure evaluation and assessment of risk trial (UK-heart). Circulation. 1998 Oct 13;98(15):1510-6. doi: 10.1161/01.cir.98.15.1510. PMID 9769304
- [Background] Myles PS, Shulman MA, Heritier S, Wallace S, McIlroy DR, McCluskey S, Sillar I, Forbes A. Validation of days at home as an outcome measure after surgery: a prospective cohort study in Australia. BMJ Open. 2017 Aug 18;7(8):e015828. doi: 10.1136/bmjopen-2017-015828. PMID 28821518
- [Background] Myles PS, Bellomo R, Corcoran T, Forbes A, Peyton P, Story D, Christophi C, Leslie K, McGuinness S, Parke R, Serpell J, Chan MTV, Painter T, McCluskey S, Minto G, Wallace S; Australian and New Zealand College of Anaesthetists Clinical Trials Network and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus Liberal Fluid Therapy for Major Abdominal Surgery. N Engl J Med. 2018 Jun 14;378(24):2263-2274. doi: 10.1056/NEJMoa1801601. Epub 2018 May 9. PMID 29742967
- [Background] Mostarda C, Castro-Filha J, Reis AD, Sevilio M Jr, Dias CJ, Silva-Filho AC, Garcia JBS, do Desterro Nascimento M, Coelho-Junior HJ, Rodrigues B. Short-term combined exercise training improves cardiorespiratory fitness and autonomic modulation in cancer patients receiving adjuvant therapy. J Exerc Rehabil. 2017 Oct 30;13(5):599-607. doi: 10.12965/jer.1735048.524. eCollection 2017 Oct. PMID 29114536
- [Background] Scott WR. Conflicting levels of rationality: regulators, managers, and professionals in the medical care sector. J Health Adm Educ. 1985 Spring;3(2 Pt 2):113-31. No abstract available. PMID 10276329
- [Background] Marinelli V, Danzi OP, Mazzi MA, Secchettin E, Tuveri M, Bonamini D, Rimondini M, Salvia R, Bassi C, Del Piccolo L. PREPARE: PreoPerative Anxiety REduction. One-Year Feasibility RCT on a Brief Psychological Intervention for Pancreatic Cancer Patients Prior to Major Surgery. Front Psychol. 2020 Mar 5;11:362. doi: 10.3389/fpsyg.2020.00362. eCollection 2020. PMID 32194490
- [Background] Lundstrom CJ, Foreman NA, Biltz G. Practices and Applications of Heart Rate Variability Monitoring in Endurance Athletes. Int J Sports Med. 2023 Jan;44(1):9-19. doi: 10.1055/a-1864-9726. Epub 2022 Jul 19. PMID 35853460
- [Background] Leite MR, Ramos EM, Kalva-Filho CA, Rodrigues FM, Freire AP, Tacao GY, de Toledo AC, Cecilio MJ, Vanderlei LC, Ramos D. Correlation between heart rate variability indexes and aerobic physiological variables in patients with COPD. Respirology. 2015 Feb;20(2):273-8. doi: 10.1111/resp.12424. Epub 2014 Nov 9. PMID 25381699
- [Background] Lavin-Perez AM, Collado-Mateo D, Mayo X, Liguori G, Humphreys L, Jimenez A. Can Exercise Reduce the Autonomic Dysfunction of Patients With Cancer and Its Survivors? A Systematic Review and Meta-Analysis. Front Psychol. 2021 Aug 24;12:712823. doi: 10.3389/fpsyg.2021.712823. eCollection 2021. PMID 34504462
- [Background] Larsen AI, Gjesdal K, Hall C, Aukrust P, Aarsland T, Dickstein K. Effect of exercise training in patients with heart failure: a pilot study on autonomic balance assessed by heart rate variability. Eur J Cardiovasc Prev Rehabil. 2004 Apr;11(2):162-7. doi: 10.1097/01.hjr.0000124214.21584.bb. PMID 15187821
- [Background] Landoni G, Lomivorotov VV, Alvaro G, Lobreglio R, Pisano A, Guarracino F, Calabro MG, Grigoryev EV, Likhvantsev VV, Salgado-Filho MF, Bianchi A, Pasyuga VV, Baiocchi M, Pappalardo F, Monaco F, Boboshko VA, Abubakirov MN, Amantea B, Lembo R, Brazzi L, Verniero L, Bertini P, Scandroglio AM, Bove T, Belletti A, Michienzi MG, Shukevich DL, Zabelina TS, Bellomo R, Zangrillo A; CHEETAH Study Group. Levosimendan for Hemodynamic Support after Cardiac Surgery. N Engl J Med. 2017 May 25;376(21):2021-2031. doi: 10.1056/NEJMoa1616325. Epub 2017 Mar 21. PMID 28320259
- [Background] Landoni G, Lomivorotov VV, Nigro Neto C, Monaco F, Pasyuga VV, Bradic N, Lembo R, Gazivoda G, Likhvantsev VV, Lei C, Lozovskiy A, Di Tomasso N, Bukamal NAR, Silva FS, Bautin AE, Ma J, Crivellari M, Farag AMGA, Uvaliev NS, Carollo C, Pieri M, Kunstyr J, Wang CY, Belletti A, Hajjar LA, Grigoryev EV, Agro FE, Riha H, El-Tahan MR, Scandroglio AM, Elnakera AM, Baiocchi M, Navalesi P, Shmyrev VA, Severi L, Hegazy MA, Crescenzi G, Ponomarev DN, Brazzi L, Arnoni R, Tarasov DG, Jovic M, Calabro MG, Bove T, Bellomo R, Zangrillo A; MYRIAD Study Group. Volatile Anesthetics versus Total Intravenous Anesthesia for Cardiac Surgery. N Engl J Med. 2019 Mar 28;380(13):1214-1225. doi: 10.1056/NEJMoa1816476. Epub 2019 Mar 19. PMID 30888743
- [Background] Lambert JE, Hayes LD, Keegan TJ, Subar DA, Gaffney CJ. The Impact of Prehabilitation on Patient Outcomes in Hepatobiliary, Colorectal, and Upper Gastrointestinal Cancer Surgery: A PRISMA-Accordant Meta-analysis. Ann Surg. 2021 Jul 1;274(1):70-77. doi: 10.1097/SLA.0000000000004527. PMID 33201129
- [Background] Kleiger RE, Miller JP, Bigger JT Jr, Moss AJ. Decreased heart rate variability and its association with increased mortality after acute myocardial infarction. Am J Cardiol. 1987 Feb 1;59(4):256-62. doi: 10.1016/0002-9149(87)90795-8. PMID 3812275
- [Background] Kemp AH, Quintana DS. The relationship between mental and physical health: insights from the study of heart rate variability. Int J Psychophysiol. 2013 Sep;89(3):288-96. doi: 10.1016/j.ijpsycho.2013.06.018. Epub 2013 Jun 22. PMID 23797149
- [Background] Kaikkonen KM, Korpelainen RI, Tulppo MP, Kaikkonen HS, Vanhala ML, Kallio MA, Keinanen-Kiukaanniemi SM, Korpelainen JT. Physical activity and aerobic fitness are positively associated with heart rate variability in obese adults. J Phys Act Health. 2014 Nov;11(8):1614-21. doi: 10.1123/jpah.2012-0405. Epub 2014 Feb 5. PMID 24508687
- [Background] Jarczok MN, Weimer K, Braun C, Williams DP, Thayer JF, Gundel HO, Balint EM. Heart rate variability in the prediction of mortality: A systematic review and meta-analysis of healthy and patient populations. Neurosci Biobehav Rev. 2022 Dec;143:104907. doi: 10.1016/j.neubiorev.2022.104907. Epub 2022 Oct 13. PMID 36243195
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Fadul N, Strasser F, Palmer JL, Yusuf SW, Guo Y, Li Z, Allo J, Bruera E. The association between autonomic dysfunction and survival in male patients with advanced cancer: a preliminary report. J Pain Symptom Manage. 2010 Feb;39(2):283-90. doi: 10.1016/j.jpainsymman.2009.06.014. PMID 20152590
- [Background] Durrand J, Singh SJ, Danjoux G. Prehabilitation. Clin Med (Lond). 2019 Nov;19(6):458-464. doi: 10.7861/clinmed.2019-0257. PMID 31732585
- [Background] Dekker JM, Crow RS, Folsom AR, Hannan PJ, Liao D, Swenne CA, Schouten EG. Low heart rate variability in a 2-minute rhythm strip predicts risk of coronary heart disease and mortality from several causes: the ARIC Study. Atherosclerosis Risk In Communities. Circulation. 2000 Sep 12;102(11):1239-44. doi: 10.1161/01.cir.102.11.1239. PMID 10982537
- [Background] De Couck M, van Brummelen D, Schallier D, De Greve J, Gidron Y. The relationship between vagal nerve activity and clinical outcomes in prostate and non-small cell lung cancer patients. Oncol Rep. 2013 Nov;30(5):2435-41. doi: 10.3892/or.2013.2725. Epub 2013 Sep 9. PMID 24026706
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Bell M, Eriksson LI, Svensson T, Hallqvist L, Granath F, Reilly J, Myles PS. Days at Home after Surgery: An Integrated and Efficient Outcome Measure for Clinical Trials and Quality Assurance. EClinicalMedicine. 2019 Apr 27;11:18-26. doi: 10.1016/j.eclinm.2019.04.011. eCollection 2019 May-Jun. PMID 31317130